CLINICAL TRIAL: NCT06733779
Title: Investigation and Analysis of the NIS Protection Level and Influencing Factors of Clinical Nurses: a Large Population Sample Survey Based on China Economic Belt
Brief Title: Investigation and Analysis of the NIS Protection Level and Influencing Factors of Clinical Nurses
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Shen Ying, associate-professor, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: K2023-192
Record Dates: First submitted 2024-12-07; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Needle Injury
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Eastern region Western region: Located in eastern region of China
  Interventions: Other: observation
- Centrel region: Located in the central region of China
  Interventions: Other: observation
- Western region: Located in western region of China
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — cross-sectional study

SUMMARY:
To investigate and analyze differences in the incidence of needle stick injuries and the influencing factors among clinical nurses in different economic regions.

The online questionnaire survey was conducted by stratified and network sampling methods. A total of 17,164 questionnaires were collected, which included demographic characteristics of nurses; knowledge, beliefs, and behaviors related to needle injury protection of nurses; hospital management, training, and assessment of "needle injury" protocols. Additionally, the knowledge, beliefs, and behaviors of nurses in needle stick injuries were compared according to the economic region, and the correlation between influencing factors was analyzed.

DETAILED DESCRIPTION:
Background: Needle stick injuries are a leading cause of occupational exposure in clinical nurse practice, with previous studies establishing that their incidence is typically lower in developed countries and affected by the local economic level. In China, significant differences in economic development levels exist between different regions. Based on the division of the economic region, this study investigated and analyzed differences in the incidence of needle stick injuries and the influencing factors among clinical nurses in different economic regions.

Methods:

The survey considered the level of economic development and regional characteristics. It included at least 5 tertiary hospitals from each provincial administrative unit, encompassing general hospitals, specialized hospitals, maternal and child health care hospitals, etc. Inclusion criteria for nurses: in-service and on-the-job clinical nurses working in tertiary hospitals holding valid nurse qualification certificates who voluntarily cooperated with the investigators. Exclusion criteria: nursing students, nursing managers, individuals taking maternity leave due to pregnancy or childbirth, refusal to participate in the survey, questionnaire completion time not meeting the minimum requirement, reverse entry selections, and incomplete responses. All study subjects were informed of the survey details in advance and signed the informed consent form before accessing the survey page.

Questionnaire This survey included a custom-made questionnaire entitled "Survey on the status of needle prick injuries in clinical nurses". It was designed by the researcher in collaboration with the experts of the clinical IV therapy team of the First Affiliated Hospital of Chongqing Medical University based on the "NSI protection expert consensus in 2018" [23] and was completed through four rounds of discussion and revisions. The expert group consisted of 13 members (including one statistical expert) distributed across five cities, seven general hospitals, and one medical college (statistical expert), among which 10 held senior titles and three held deputy senior titles. The questionnaire was reviewed by via four rounds of expert consultations from seven hospitals. Considering the influence of regional cultural differences in written expression, 268 pilot questionnaires were initially conducted in Chongqing (Western region), Guangdong (Southern region), and Hebei (Northern region) to further refine language and content. Finally, the questionnaire comprised three sections: 1. demographic characteristics of nurses, including region, hospital name, department name, age, years of experience, nursing role, nurse title, educational level, etc.; 2. Knowledge, belief, and behavior of nurses regarding NSI protection; 3. Hospital management, training, and assessment of the implementation of "NSI protection". The Kronbuck coefficient of the knowledge, belief, and behavior questionnaire was 0.789.

Based on the population data of each provincial administrative unit in 2021 [24], a stratified sampling method was employed based on a ratio of 1/100,000 population for each unit. The online questionnaire survey was distributed through an online survey software (Questionnaire Star) combined with an online sampling method. China Nursing Association is the only national nursing association organization for Nurses in China, with the Hospital Infection Management Committee of the Chinese Nursing Society being a subdivision of the organization. Its members are distributed in 28 provincial administrative units across the country, with over 800 members and 130 nursing department directors. This survey was officially published by the Hospital Infection Management Committee of the Chinese Nursing Society. Following approval of the survey notification information and questionnaire by the committee, the committee informed the liaison officers of the national hospital infection management committee to inform the head nurses of the hospital through the official WeChat working group, who in turn shared the questionnaire in the WeChat working groups of the department nurses. The notice asked the head nurse to emphasize the principle of voluntariness to the investigation object when sharing the questionnaire.

After the completion of the round of the survey, the researchers compiled completed statistics for each province and contacted liaison officers of local hospitals for the provinces that failed to meet the standards to launch a new round of data collection in the hospital. The survey was conducted from 8:00 on November 9, 2022, to 20:00 on February 16, 2023. Each round of surveys lasted 1 week.

Quality control When transcribing the questionnaire into an electronic format, two persons were accountable for logical consistency. To exclude invalid responses, a screening page was set, option quotas were established, the time for responses was controlled, and the answer input areas were restricted. Additionally, restrictions were imposed to allow login exclusively via WeChat, with each IP address and physical address limited to a single submission.

Data collection In order to ensure the integrity and reliability of the questionnaire, an informed consent page and explanation page were set up to detail the purpose and significance of the survey, as well as participant requirements, instructions, etc. The respondent could proceed with the questionnaire by selecting "agree to conduct the survey". The features of the questionnaire were as follows: 1. Set the questionnaire topic as the required topic; 2. requiring complete responses, with incomplete submissions being automatically rejected; 3. Setting the minimum time of completion to 5'20" according to the pre-survey, with submissions below this threshold automatically classified as invalid. A total of 17,164 questionnaires were collected, including 15,274 valid questionnaires, yielding an effective response rate of 89.89%.

Statistical method Categorical data were described as frequencies and rates, and group comparisons were performed using the chi-square test, with p-values adjusted using the S method for post-hoc pairwise comparisons. Measurement data following a normal distribution were presented mean ± standard deviation and compared using the two independent samples t-test or ANOVA, and post-hoc pairwise comparisons were conducted using the SNK-q test. Variables with P <0.05 in the univariate analysis were incorporated in a multivariate linear regression model to identify factors influencing the total score of the respondents and were screened using the stepwise selection method.

Variables with P <0.05 in the univariate analysis were incorporated in a multivariate linear regression model to identify factors influencing the total score of the respondents and were screened using the stepwise selection method with inclusion criteria for P <0.05 and exclusion for P ≥0.05.

The multiple mediation effect model was utilized to elucidate the association between economic regions and needle stick injury and to quantify the indirect and direct associations between economic regions through needle stick injury-related management, assessment, and training as mediating variables. In the present study, considering that multiple mediating variables were dichotomous variables, the indirect effects were challenging to directly measure. Therefore, the indirect effect size was quantified by the percentage of mediation (percentage mediated, PM), formula 1 minus the ratio of the direct effect (Direct effect, DE) to the total effect (Total effect, TE) multiplied by 100%: PM= (1-DE/TE) x 100%. This calculation was implemented using a partial macro program.

All statistical analyses were performed using SAS 9.4. P <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

- cetificated nurse; voluntarily cooperated with the investigators;

Exclusion Criteria:

- nursing students,; nursing managers; individuals taking maternity leave due to pregnancy or childbirth; refusal to participate in the survey, questionnaire completion time not meeting the minimum requirement; reverse entry selections; incomplete responses.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: in-service and on-the-job clinical nurses working in tertiary hospitals
Sampling Method: Non-Probability Sample
Enrollment: 17164 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
differences in the incidence of needle stick injuries and the influencing factors among clinical nurses in different economic regions. | up to 12 weeks.
  to analyze the incidence rate in different regions and ralated influencing factors.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Shen, M.D, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- the First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided